CLINICAL TRIAL: NCT02232919
Title: Hypothalamus Deep Brain Stimulation for Human Morbid Obesity: Feasibility Trial
Brief Title: Deep Brain Stimulation for Human Morbid Obesity
Acronym: BLESS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230/2012
Record Dates: First submitted 2014-08-21; First posted 2014-09-05 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Obesity | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): The design of this translation trial is a single-center, single cohort, open-label and non-masked study. The aim is to evaluate tolerability of chronic low-frequency electrical stimulation of the VMH, while achieving weight loss in morbidly obese subjects. The subjects must have a body-mass index [BMI] greater than 40, and no obesity co-morbidities, such as diabetes or cardiopulmonary abnormalities. Up to six subjects will be implanted in this protocol.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — If subjects qualify with respect to protocol requirements, the Medtronic Activa system will be implanted with the leads placed bilaterally in the VMH.
  Adjustment of DBS parameters at the three months visit will be performed to improve efficacy when the goal of 3% body weight loss mark was not achieved during this period of continuous stimulation. Subjects will be seen monthly after discharge throughout the study period. At visits, safety will be assessed through blood/urine tests, blood pressure measurements, verbal interviews with the subjects and family, quarterly formal psychiatric tests as well as QOL scales.
  The determination of efficacy will be the within-group percent change in weight at the end of the DBS treatment period compared to baseline.

SUMMARY:
The burden of morbid obesity to the circulatory, endocrine, and locomotor systems, as well as the psychological effects and related health-care costs, are well established in the medical literature. Lifestyle and dietary patterns remain critical factors modulating long-term weight control of morbidly obese individuals (bodymass index ≥ 40). Various dietary, pharmacological, and behavioral interventions have largely failed as therapies, often necessitating surgery as the last treatment option. Long term results of bariatric surgery suggest that sustained and substantial weight loss can decrease morbidity related to obesity secondary complications such as diabetes type 2 and cancers, enhancing the role of surgery for morbidly obese subjects. However the adverse effects of bariatric surgery are considerable and impact on quality of life. Its long-term failure rates and complications call for novel and effective long-term therapies, such as neurosurgical interventions.

The investigators now propose to enhance our targeting capabilities in a feasibility study of low frequency electrical stimulation using VMH-DBS (ventromedial hypothalamic) in six morbidly obese patients. After successful targeting, DBS stimulation parameters will be systematically evaluated and individually optimized at three-month intervals over a one-year stimulation period. Detailed recording of side effects, weight changes, food intake patterns, metabolic changes, and behavioral evaluations will be obtained throughout the study.

DETAILED DESCRIPTION:
Neuromodulation of metabolism and feeding behavior is at hand using modern systems of deep brain stimulation (DBS). It constitutes a minimally invasive approach for these challenging patients. The surgical procedure is reversible and proven to have acceptable side effects in the frail population of Parkinson's disease patients [Gorgulho, Hemorrhage and Infection]. Improvement of functional stereotactic surgery methods is necessary however to the challenge of implanting DBS electrodes in the hypothalamus. Recently, a case report of a patient with DBS implanted in the hypothalamus for treatment of morbid obesity who reported side effects related to memory appeared in the literature. The authors used the side effect findings to suggest the location of their implant as a site for treatment of Alzheimer's disease. This illustrates the need of betterment of our techniques of targeting in DBS surgery, especially for targets located in highly functional structures, such as the hypothalamus.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index [BMI] >40 kg/m2. BMI definition = weight [Kg] / height [m]2
2. Failed diet, exercise, behavior, and pharmacotherapy to control body weight.

Exclusion Criteria:

1. Cancer requiring treatment in the past five years, with the exception of cancers which have been cured or, in the opinion of the investigator, carry a good prognosis [for example, non melanoma skin cancer].
2. Infectious disease [e.g., HIV or active tuberculosis].
3. Cardiovascular disease:

   i. Hospitalization for treatment of heart disease in the past 6 months. ii. New York Heart Association Functional Class >2. iii. Left bundle branch block on EKG. iv. Third degree atrioventricular block on EKG. v. Uncontrolled hypertension [average systolic blood pressure of >160 mmHg or diastolic blood pressure >95 mmHg on both screening visits].

   vi. Pulse rate >95 beats per minute on both screening visits. vii. Total serum cholesterol >300 mg/dL. viii. Stroke or transient ischemic attack in the past 6 months.
4. Gastrointestinal disease:

   i. Chronic hepatitis or cirrhosis. ii. Episode of alcoholic hepatitis or alcoholic pancreatitis. iii. Inflammatory bowel disease requiring treatment in the past year. iv. Recent or significant abdominal surgery [e.g., gastrectomy or gastric bypass].
5. Renal disease:

   i. Serum creatinine >1.5 mg/dL. ii. Urine protein>2+ on dipstick at screening and or 24-hour urinary excretion of albumin>500 mg/day.
6. Lung disease:

   i. Chronic obstructive airway disease or asthma requiring daily therapy. ii. Use of home oxygen.
7. Endocrine disease:

   i. Diabetes mellitus. ii. Hyperlipidemia with triacylglycerol >500 mg/dL. iii. Hypothyroidism, hyperthyroidism. iv. Hypopituitarism. v. Hypogonadism.
8. Psychological Disease:

   i. Major clinical depression. ii. Active psychiatric disorders. iii. Schizophrenia.
9. Hematology i. Anemia [hematocrit <36.0%]. ii. Bleeding disorders, thrombocytopenia, thrombocytosis.
10. Conditions or behaviors likely to affect the conduct of the study:

    i. Unable or unwilling to give informed consent. ii. Unable to communicate with the clinic staff. iii. Weight loss >10% in the past 6 months. iv. Unable to walk 0.25 miles in 10 minutes. v. Behavioral disorder which, in the opinion of the investigator, would impede conduct of the study.

    vi. Excessive alcohol intake, use of illicit drugs.
11. Conditions related to medications:

    i. Psychoactive agents. ii. Monoamine oxidase inhibitors [e.g., phenelzine, procarbazine, selegiline, furazolidone].

    iii. Antidepressants [e.g., lithium, fluoxetine, sertraline, nefazodone, paroxetine, venlafaxine].

    iv. Any other medication that, in the opinion of the investigator, may pose harm to the subject.
12. Seizure disorders.
13. Receiving anticoagulation medications or likely to need anticoagulation in the foreseeable future.
14. Subject is not a surgical candidate.
15. Lack of social support.
16. Inability to comply with testing and follow-up visit requirements defined by the Study Protocol.
17. Subject has another implanted device or metallic object [e.g., cardiac demand pacemakers, aneurysm clips, cochlear implant, spinal cord stimulator, etc].
18. Subject has a medical condition that might require repeat MRIs.
19. Subject has concurrent infection.
20. Subject has any medical condition contraindicating a chronically implanted device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Identification of possible adverse events related to stimulation of the VMH | 12 months
  To identify potential side effects of continuous electrical stimulation of the VMH and optimize electrophysiological parameters to avoid these side effects in morbidly obese subjects.

SECONDARY OUTCOMES:
Body Weight | 12 months
  To determine if continuous VMH-DBS will lead to weight loss in morbidly obese subjects. Baseline measurements of body weight [kg, lb] will be recorded on 3 different occasions prior to DBS implantation. The baseline weight will be considered the arithmetic mean of these measurements. Body weight will be recorded at every follow-up visit.
Body Composition | 12 months
  To determine if continuous electrical stimulation of the VMH will lead to changes in body composition. Measurements of body composition will be evaluated by Dual-Energy Xray Absorptiometry [DEXA] at baseline and at 3 month intervals.
Food Intake. | 12 months
  To determine if VMH-DBS will cause decreased food intake. Subjects will complete a questionnaire during the monthly visit assisted by the study coordinator. Data reflecting food quality and quantity will be compiled for analysis and correlation with the other parameters obtained in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gorgulho, MD, MSc, Study Chair — HOSPITAL DO CORAÇÃO; Antonio De Salles, M.D., Ph.D., Study Chair — HOSPITAL DO CORAÇÃO; Otavio Berwanger, MD,PhD, Study Director — HOSPITAL DO CORAÇÃO
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] De Salles AAF, Barbosa DAN, Fernandes F, Abucham J, Nazato DM, Oliveira JD, Cury A, Biasi A, Rossi R, Lasagno C, Bueno PT, Santos RHN, Damiani LP, Gorgulho AA. An Open-Label Clinical Trial of Hypothalamic Deep Brain Stimulation for Human Morbid Obesity: BLESS Study Protocol. Neurosurgery. 2018 Oct 1;83(4):800-809. doi: 10.1093/neuros/nyy024. PMID 29538761